CLINICAL TRIAL: NCT01343134
Title: Anatomical and Functional Macular Changes in Retinal Detachment
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Pr Catherine Creuzot-Garcher, Ophthalmology department
Other Study IDs: Marie Pierre 01
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-01

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Retina; Rhegmatogenous retinal detachment; Macular detachment; Spectral domain OCT; Microperimetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Retinal detachment cohort
  Interventions: Device: Measure the outer retina by spectral domain optical coherence tomography (HRA Spectralis; Heidelberg), and microperimetry (OPKO Instruments)

INTERVENTIONS:
Device: Measure the outer retina by spectral domain optical coherence tomography (HRA Spectralis; Heidelberg), and microperimetry (OPKO Instruments) — Measure the thickness of the outer retina by spectral domain optical coherence tomography (HRA Spectralis; Heidelberg)and perform central microperimetry using new OPKO Instruments OCT.

SUMMARY:
The purpose of this study is to evaluate the correlation between morphologic changes in the outer retina and visual function after successful repair of rhegmatogenous retinal detachment with macula off.

ELIGIBILITY:
Inclusion Criteria:

* Rhegmatogenous retinal detachment

Exclusion Criteria:

* Epiretinal membrane

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with successful repair of rhegmatogenous retinal detachment after macula off and minimum 6 month follow-up after surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Creuzot-Garcher, MD;PhD, Study Director — Ophthalmology department CHU Dijon; Marie Pierre Delolme, MD, Principal Investigator — Ophthalmology Department CHU Dijon
Locations (1):
- Ophthalmology Department CHU Dijon, Dijon, Burgundy, France